CLINICAL TRIAL: NCT02386644
Title: Premature Rupture of Membranes Assessment Via Transperineal Ultrasonography as an Alternative to Speculum Examinations
Brief Title: Transperineal Ultrasonography and Premature Rupture of Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Erkan Kalafat, Medical Doctor, Ankara University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2015-02-21; First posted 2015-03-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Preterm Premature Rupture of the Membranes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Suspected Membrane Rupture Arm (Experimental): Women with suspected membrane rupture will be subject to following interventions; Ultrasound amniotic fluid index measurement, ultrasound transperineal assessment, nitrazine test, speculum examination, PAMG-1 Immunoassay
  Interventions: Other: PAMG-1 Immunoassay; Device: Ultrasound transperineal assessment; Device: Ultrasound amniotic fluid index measurement; Other: Speculum examination; Other: Nitrazine test

INTERVENTIONS:
Other: PAMG-1 Immunoassay — Immunoassay for presence of placental alfa microglobulin-1(PAMG) in vaginal fluids.
  Other Names: AmniSure test (AmniSure International LLC, Boston, USA)
Device: Ultrasound transperineal assessment — Transperineal ultrasound assessment of vaginal canal for pooling of amniotic fluid.
Device: Ultrasound amniotic fluid index measurement — Calculation of amniotic fluid index in millimetres via ultrasonography by measuring four deepest pockets in four quadrants.
Other: Speculum examination — Sterile speculum examination to evaluate vaginal pooling of amniotic fluid pooling.
Other: Nitrazine test — To assess acid , alkaline status of pooled fluid in vagina.

SUMMARY:
This study's aim is to evaluate diagnostic accuracy of transperineal ultrasound assessment compared with speculum examination, nitrazine and placental micro globulin-1 tests.

DETAILED DESCRIPTION:
Women with early and late preterm pregnancies with a complaint of fluid leakage are enrolled in the study. Prior to speculum examination, sagittal view of the birth canal and transverse view of cervix and fornices are obtained with transperineal technique and images are stored. Then speculum examination for pooling, nitrazine test and placental microglobulin-1 tests are performed and results are recorded. Ultrasound images are analysed by an observer blind to physical examination findings. Hypoechogenic fluid appearance of adequate size around the cervix and in the fornices are considered positive. Placental microglobulin-1 test is used as reference. Sensitivity and specificity values are calculated for each test.

ELIGIBILITY:
Inclusion Criteria:

* Women with early and late preterm pregnancies, (i.e., women above 24th and below 37th week of gestation)
* Pregnant women with a complaint of fluid leakage

Exclusion Criteria:

* Women with term pregnancies (i.e., women above 37th week of gestation)
* Women with unviable pregnancies (i.e., women below 24th week of gestation)
* Women in active labor (i.e., cervical dilatation above 4cm during admission)
* Women with vaginal bleeding

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
True positive and negative percent agreement between transperineal assessment and PAMG-1 immunoassay as reference test. | Up to 3 months
  True positive rate and true negative rate of transperineal assessment will be calculated in percentages compared to PAMG-1 immunoassay as reference test.

CONTACTS AND LOCATIONS:
Overall Officials: Acar F Koc, Professor, Study Director — Department of Obstetrics and Gynecology, Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Department of Obstetrics and Gynecology, Ankara, Turkey (Türkiye)